CLINICAL TRIAL: NCT05068388
Title: A Phase 2, Randomized, Double-blinded, Placebo-controlled, Dose-Response Study of Oral (Z)-Endoxifen in Premenopausal Women With Measurable Breast Density
Brief Title: Effect of Oral (Z)-Endoxifen in Premenopausal Women With Measurable Breast Density
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Atossa Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATOS-016R
Record Dates: First submitted 2021-09-27; First posted 2021-10-05 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Breast Density
MeSH Terms: interventions — 4-hydroxy-N-desmethyltamoxifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): oral capsule
  Interventions: Drug: Placebo
- 1 mg (Z)-endoxifen (Experimental): oral capsule
  Interventions: Drug: Z-Endoxifen
- 2 mg (Z)-endoxifen (Experimental): oral capsule
  Interventions: Drug: Z-Endoxifen

INTERVENTIONS:
Drug: Z-Endoxifen — Z-Endoxifen
  Arms: 1 mg (Z)-endoxifen; 2 mg (Z)-endoxifen
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blinded, placebo-controlled dose-response efficacy study of oral (Z)-endoxifen in premenopausal women with measurable breast density. There will be 5 in-clinic visits (Screening, Day 1, Months 1, 3 and 6) and 3 self-report visits (Months 2, 4 and 5). Standard of care mammograms will be used for the screening mammogram as well as the 24-month follow up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal women (defined as having at least one menstruation during the prior 12 months; women with an intrauterine device are considered premenopausal if <52 years)
2. Women of childbearing potential using a highly effective method of birth control* throughout the study period and willing to comply with monthly pregnancy testing
3. Screening mammogram performed within 3 month of study inclusion
4. Mammographic density assessed as BI-RADS® score B, C, or D
5. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects

Exclusion Criteria:

1. Mammographic BI-RADS® malignancy code ≥3 at baseline mammography
2. Any previous diagnosis of breast cancer, including carcinoma in situ, or any other cancer (non-melanoma skin cancer and in situ cancer of the cervix are not exclusion criteria)
3. A history of breast surgery, e.g., reduction or enlargement, which might affect mammographic density measurements
4. Current medical conditions:

   1. APC (activated protein C) resistance, an inherited coagulation disorder
   2. Systolic pressure higher than 160 mm Hg or diastolic higher than 100 mm Hg
   3. Cataract(s)
   4. Uncontrolled diabetes (defined as HbA1c >50 mmol/mol)
   5. Abnormal lab values deemed clinically significant by Investigator
5. BMI > 30
6. Women who have an increased risk of venous thrombosis due to immobilization, e.g., using wheelchair
7. Agents that have the potential to decrease endoxifen levels through increased metabolic clearance:

   1. Certain anti-epileptic therapies (carbamazepine, fenytoin, fenobarbital, lamotrigine)
   2. Certain antibiotics (rifamycins)
   3. St John's wort (in Swedish: johannesört)
   4. Certain HIV medications (efavirenz, ritonavir)
8. Lactating, pregnant, or plan to become pregnant in the next year
9. History of thromboembolic disease such as embolus, deep vein thrombosis, stroke, TIA (transient ischemic attack) or myocardial infarction
10. Allergy to endoxifen or any of its components
11. Previous treatment with an anti-oestrogen, including experimental drug studies (e.g., Karma CREME, Karisma-1 or Karisma-2)
12. Prescribed and regular use of anticoagulants (defined as substances included in group B01A in the ATC-system)
13. Participation in another investigational clinical trial in the last 6 months
14. Not willing or able to understand the study information and/or informed consent

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — having at least one menstruation during the prior 12 months; women with an intrauterine device are considered premenopausal if <52 years
Enrollment: 240 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2024-08-28 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of mammographic density area (cm2) assessed by iCAD® software | 6 months
  Change from baseline

SECONDARY OUTCOMES:
Change of mammographic density area (cm2) assessed by iCAD® software | 3 months
  Change from baseline
Change of mammographic density area (cm2) assessed by Stratus software | 6 months
  Change from baseline
Change of mammographic density area (cm2) assessed by Stratus software | 3 months
  Change from baseline
Change from baseline responses to the Breast Cancer Prevention Trial Eight Symptom Scale (BESS) | 6 months
  5-point Likert-type scale
Comparison of adverse events | 6 months
  assessment of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Steven Quay, MD, Study Director — Atossa Therapeutics, Inc.; Per Hall, MD, Principal Investigator — Södersjukhuset, Stockholm, Sweden
Locations (1):
- Karma Study Centre, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No